CLINICAL TRIAL: NCT02526498
Title: TRI-fraction Radiotherapy Utilized to Minimize Patient Hospital Trips : A Phase II Trial (TRIUMPH-T Trial)
Brief Title: Accelerated Partial Breast Radiation Therapy Using High-Dose Rate Brachytherapy in Treating Patients With Early Stage Breast Cancer After Surgery
Acronym: TRIUMPH-T
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Rutgers Cancer Institute of New Jersey (Other); Cianna Medical, Inc. (Industry); Elekta Limited (Industry)
Responsible Party: Principal Investigator, Bruce G Haffty, Principal Investigator, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 041404; NCI-2015-01156 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro20150001297 (Other: IRB Number); Pro20150001297 (Other: Rutgers Cancer Institute of New Jersey)
Record Dates: First submitted 2015-08-04; First posted 2015-08-18 (Estimated); Results first posted 2022-08-16 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-04

CONDITIONS: Ductal Breast Carcinoma In Situ; Estrogen Receptor Positive; Invasive Breast Carcinoma; Progesterone Receptor Positive; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (APBI using HDR brachytherapy) (Experimental): Within 1-5 days after balloon placement, patients undergo APBI using HDR brachytherapy over 15-60 minutes for 2-3 days.
  Interventions: Radiation: Accelerated Partial Breast Irradiation; Radiation: High-Dose Rate Brachytherapy; Other: Questionnaire Administration

INTERVENTIONS:
Radiation: Accelerated Partial Breast Irradiation — Undergo accelerated partial breast irradiation (APBI) using high-dose rate (HDR) brachytherapy
  Other Names: APBI
Radiation: High-Dose Rate Brachytherapy — Undergo APBI using HDR brachytherapy
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well accelerated partial breast irradiation (APBI) using high-dose rate (HDR) brachytherapy works in treating patients with breast cancer that has not spread beyond the breast or the axillary lymph nodes (early-stage) after surgery. Radiation therapy uses a type of energy to kill cancer cells and shrink tumors. Brachytherapy is a type of internal radiation therapy that provides radiation inside the breast to any remaining tumor cells next to the space where the tumor was removed, and is given over a shorter amount of time than standard radiation therapy. Giving accelerated partial breast irradiation (APBI) using high-dose rate (HDR) brachytherapy may reduce the overall time that radiation is delivered to the tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the toxicity rate with shorter courses of accelerated partial breast irradiation (APBI) delivered with a breast brachytherapy applicator.

SECONDARY OBJECTIVES:

I. To determine the 3-year actuarial local control rate with abbreviated accelerated partial breast irradiation (APBI).

II. To assess the rate of excellent or good cosmesis at 2-years after shorter courses of APBI and to identify co-variants associated with and predictive of poor cosmetic outcome in women treated with an overnight treatment course of APBI.

OUTLINE:

Within 1-5 days after balloon placement, patients undergo accelerated partial breast irradiation (APBI) using high-dose rate (HDR) brachytherapy over 15-60 minutes for 2-3 days.

After completion of study treatment, patients are followed up at 2-8 weeks and then at least annually for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Must sign informed consent
* Surgical treatment of the breast must have been lumpectomy; the margins of the resected specimen must be histologically free of tumor (negative surgical margins per National Surgical Adjuvant Breast and Bowel Project [NSABP] criteria)
* On histologic examination, the tumor must be ductal carcinoma in situ (DCIS) and/or invasive breast carcinoma
* For patients with invasive breast cancer, an axillary staging procedure must be performed (either sentinel node biopsy [SNB] alone or axillary dissection [with a minimum of six axillary nodes removed], and the axillary node[s] must be pathologically negative); patients over 70 with estrogen receptor positive (ER+) tumors no greater than 2 cm do not require axillary evaluation, but MUST be clinically node negative on examination and all available imaging (clinical N0)
* The T stage must be Tis, T1, or T2; if T2, the tumor must be =< 3.0 cm in maximum diameter
* Estrogen receptor positive tumor and/or progesterone receptor positive tumor

Exclusion Criteria:

* Pregnant or breast-feeding
* Active collagen-vascular disease
* Paget's disease of the breast
* Prior history of DCIS or invasive breast cancer
* Prior breast or thoracic radiation therapy (RT) for any condition
* Multicentric carcinoma (DCIS or invasive)
* Synchronous bilateral invasive or non-invasive breast cancer
* Surgical margins that cannot be microscopically assessed or that are positive
* Positive axillary node(s)
* T stage of T2 with the tumor > 3 cm in maximum diameter or a T stage >= 3
* Estrogen receptor negative and progesterone receptor negative tumor
* Any of the dosimetric treatment criteria as defined have not been met; patients who become ineligible due to inability to meet dosimetric criteria should not receive treatment as defined in this protocol and will come off the study; any subsequent adjuvant radiation will be delivered at the discretion of the treating physician

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Haffty, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (10):
- United States (10):
  - Arizona Breast Cancer, Gilbert, Arizona
  - University of California, San Diego, La Jolla, California
  - William Beaumont Hospital Research Institute, Royal Oak, Michigan
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - 21st Centry Oncolgy, Yonkers, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Huntsman Cancer Hospital, University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan AJ, Chen PY, Yashar C, Poppe MM, Li L, Abou Yehia Z, Vicini FA, Moore D, Dale R, Arthur D, Shah C, Haffty BG, Kuske R. Three-Fraction Accelerated Partial Breast Irradiation (APBI) Delivered With Brachytherapy Applicators Is Feasible and Safe: First Results From the TRIUMPH-T Trial. Int J Radiat Oncol Biol Phys. 2019 May 1;104(1):67-74. doi: 10.1016/j.ijrobp.2018.12.050. Epub 2019 Jan 4. PMID 30611839

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (APBI Using HDR Brachytherapy)
Started | 200
Completed | 200
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (APBI Using HDR Brachytherapy)
Number analyzed (Participants) | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 65
  >=65 years | 135
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 189
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 185
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 200

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Greater Than Grade 2 Serious Toxicity Rate, Defined as Toxicity Greater Than Grade 2 Using Common Terminology Criteria for Adverse Events Version 4.0 Criteria
Description: Measured by the data collected for toxicity and cosmesis as dichotomous variables. This will be assessed by physical examination at each follow-up visit. To be scored as a serious toxicity counting toward the primary endpoint, the toxicity must have a "probable" or "definite" attribution to the study treatment.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (APBI Using HDR Brachytherapy)
Number analyzed (Participants) | 200
Participants | 200

2. Secondary Outcome: Local Control Rate, Assessed by Physical Examination
Description: The association of variables with local regional failure times will be investigated by fitting a parametric model and examining the significance of the parameter estimates. Nonparametric estimates of the survival or recurrence-free distributions or recurrence (failure) distribution will be obtained by life table methods.
Time Frame: 3 years
Population: Data not collected.
Arm/Group | Treatment (APBI Using HDR Brachytherapy)
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Good/Excellent Cosmetic Results, Using the Harvard Cosmesis Scale
Description: Descriptive statistics reported.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (APBI Using HDR Brachytherapy)
Number analyzed (Participants) | 182
Participants | 177

4. Secondary Outcome: Local Control Rate, Assessed by Mammography
Description: Assessed using the Kaplan-Meier method. The association of variables with local regional failure times will be investigated by fitting a parametric model and examining the significance of the parameter estimates. Nonparametric estimates of the survival or recurrence-free distributions or recurrence (failure) distribution will be obtained by life table methods. Tests will be declared statistically significant if the calculated P-value was =< 0.05. All tests appear as 2-sided P-values.
Time Frame: 3 years
Population: Data not collected.
Arm/Group | Treatment (APBI Using HDR Brachytherapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of two years.
Arm/Group | Treatment (APBI Using HDR Brachytherapy)
All-Cause Mortality (participants affected / at risk) | 0/200
Serious Adverse Events (participants affected / at risk) | 0/200
Other Adverse Events (participants affected / at risk) | 165/200
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (APBI Using HDR Brachytherapy) (N=200)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 44 (58)
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 29 (37)
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 19 (19)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 39 (42)
Dermatitis radiation (Skin and subcutaneous tissue disorders) | 29 (32)
Seroma (Skin and subcutaneous tissue disorders) | 11 (11)
Reproductive system and breast disorder (Reproductive system and breast disorders) | 35 (41)
Breast Pain (General disorders) | 30 (38)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT02526498/Prot_SAP_ICF_000.pdf